CLINICAL TRIAL: NCT01663753
Title: Diagnostic Performance of 18F-FDG-PET and Diffusion-weighted MRI in the Assessment of Stage IB to IIB2 Cervical Squamous-cell Carcinoma Response to Concomitant Radiochemotherapy and Brachytherapy
Acronym: ERRICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011.670/13
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Cancer of the Uterine Cervix
Keywords: 2-fluoro-2-deoxy-d-glucose-positron emission tomography; Positron emission tomography; Magnetic resonance imaging; Diffusion weighted MRI; Squamous-cell cervical carcinoma; Sensitivity
MeSH Terms: conditions — Uterine Cervical Neoplasms; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-FDG-PET (Experimental): The 18F-FDG-PET will be performed 8 weeks following completion of brachytherapy (date of inclusion)
  Interventions: Device: 18F-FDG-PET

INTERVENTIONS:
Device: 18F-FDG-PET

SUMMARY:
Rationale: The benefit-risk ratio of surgery following concomitant radiochemotherapy and brachytherapy remains to be defined in cervical squamous-cell carcinoma (SCC) treatment. Scarce studies evaluated the interest of 18F-FDG-PET and MRI in the assessment of response to treatment before surgery. A positive predictive value of 75% was found in a small study making 18F-FDG-PET a promising tool to assess tumor response and guide surgical approach. Diffusion-weighted MRI was also described as an early and sensitive indicator in other diseases.

Objectives: The main objective of this study is to evaluate the sensitivity of 18F-FDG-PET in the assessment of cervical cancer response to radiochemotherapy and brachytherapy. Secondary objectives focus on 18F-FDG-PET specificity and likehood ratios as well as diffusion-weighted MRI diagnostic performances.

Method: We will conduct a prospective cohort study of 148 women with a stage IB to IIB2 cervical SCC recruited over 2.5 years in 24 centers in France. Each patient will undergo a 18F-FDG-PET and a diffusion-weighted MRI before surgery and 8 weeks after completion of the brachytherapy. The total follow-up duration (study participation) of patients will be 11 weeks : inclusion after completion of radiochemotherapy and brachytherapy, 8 weeks until 18F-FDG-PET and diffusion-weighted MRI, and 3 weeks until surgery.

Expected results: 18F-FDG-PET and diffusion-weighted MRI could constitute a reliable tool to assess response to radiochemotherapy and brachytherapy in cervical SCC treatment. If so it could improve clinical practices and be helpful to decide whether the patient needs surgery or not after radiochemotherapy and brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years of age or older
* Biopsy-confirmed cervical squamous-cell carcinomas
* Stage IB2, IIA ou IIB according to the FIGO staging of cervical carcinomas
* No spread to lumbo-aortic lymph nodes
* No prior pelvic radiotherapy
* No prior cancer treatment
* WHO Performance status less than or equal to 1
* Beneficiary of a health insurance
* Must provide her signed and informed consent

Exclusion Criteria:

* Reccurent or Metastasized cancer
* History of uncontrolled cancer, or any cancer treated for less than 5 years (except basal cell carcinomas)
* Any contraindication to MRI
* Know hypersensitivity to Gadolinium, 18F-FDG or one of the excipients
* Pregnant or breast feeding patients
* Participation in any other clinical trial that could interfere with the study results
* Any geographical, social or psychical reasons that could prohibit the ability to return for follow-up assessment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity of 18F-FDG-PET in the assessment of stage IB to IIB2 cervical squamous-cell carcinoma response to concomitant radiochemotherapy and brachytherapy | 8 weeks
  A centralized review will be carried out by 2 independant reviewers, additionally to the initial interpretation. The gold-standard to evaluate tumoral response to radiochemotherapy and brachytherapy will be the anatomopathologic analysis of the hysterectomy piece after surgery. The18F-FDG-PET will be performed 8 weeks following completion of brachytherapy (date of inclusion)and surgery will be performed within 3 weeks after the 18F-FDG-PET.

SECONDARY OUTCOMES:
Specificity and likehood ratios of 18F-FDG-PET in the assessment of stage IB to IIB2 cervical squamous-cell carcinoma response to concomitant radiochemotherapy and brachytherapy | 8 weeks
Diagnostic performances of diffusion-wheighed MRI in the assessment of stage IB to IIB2 cervical squamous-cell carcinoma response to concomitant radiochemotherapy and brachytherapy | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GOLFIER François, MD, PhD, Principal Investigator — Centre Hospitalier Lyon Sud, Hospices Civils de Lyon
Locations (24):
- France (24):
  - Service de Médecine Nucléaire, Institut de cancérologie de l'Ouest - Site Paul Papin, Angers
  - Service Gynécologie Obstétrique, Hôpital Pellegrin, CHU Bordeaux, Bordeaux
  - Service de Gynécologie, Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Bron
  - Service de Chirurgie Oncologique, Centre de Lutte Contre le Cancer Georges-François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Service de Gynécologie Obstétrique, Hôpital de la Croix-Rousse, Hospices Civils de Lyon, Lyon
  - Service de Gynécologie Obstétrique, Hôpital Nord, Marseille
  - Service de Chirurgie Gynécologique, Hôpital Arnaud de Villeneuve, Montpellier
  - Service de Radiothérapie, C.R.L.C. Val d'Aurelle, Montpellier
  - Service de Gynécologie, Hôpital Archet II, Nice
  - Service de Gynécologie, Hôpital Européen Georges Pompidou, APHP, Paris
  - Service de Gynécologie Obstétrique, Hôpital Tenon, APHP, Paris
  - Service de Chirurgie Gynécologique, Institut Curie, Paris
  - Service de Gynécologie Obstétrique, Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite
  - Service de Gynécologie Obstétrique, CHU la Milétrie, Poitiers
  - Service de Gynécologie Obstétrique, CHU Anne de Bretagne Hôpital Sud, Rennes
  - Département des Radiations, Centre Eugène Marquis, Rennes
  - Service de Chirurgie, Centre Henri Becquerel, Rouen
  - Service de Chirurgie Gynécologique, Institut Curie - Hôpital René Huguenin, Saint-Cloud
  - Service de Gynécologie Obstétrique, CHU St-Etienne, Saint-Etienne
  - Servce de Médecine Nucléaire, Centre René Gauducheau, CRLCC Nantes Atlantique, Saint-Herblain
  - Département de Radiothérapie, Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Service de Médecine Nucléaire, Hôpital Brabois, Vandœuvre-lès-Nancy
  - Service de Chirurgie Oncologique, Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy